CLINICAL TRIAL: NCT04377451
Title: Metformin as Adjunctive Therapy in Overweight and Obese Patients With Dengue: an Open-label Safety and Tolerability Trial
Brief Title: Metformin in Dengue With Obesity
Acronym: MeDO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 56DX
Record Dates: First submitted 2020-04-22; First posted 2020-05-06 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Dengue; Viral Infection; Metformin; Anti-inflammatory Agents; Obesity; Overweight
Keywords: Dengue; Obesity; Metformin; Vietnam
MeSH Terms: conditions — Dengue; Virus Diseases; Obesity; Overweight | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This is an open-label, two-phase dose escalation trial of metformin in overweight/obese patients with dengue compared to standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): The control group will be formed of 60 overweight or obese dengue patients receiving standard of care
- Intervention arm (Experimental): Two cohorts receive a 5-day course of metformin treatment. In the initial phase (cohort 1), 5 young adults and 5 children (age <16) will receive a low dose of metformin. In the second phase (cohort 2), 25 adult and 25 paediatric patients will receive a weight-based dose of metformin.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — The trial will be conducted in two phases, with a dose escalation of metformin. Metformin dosing will begin at 500mg (children) and 850mg (adults) once daily for 5 days in cohort 1.
  Cohort 2 will be received weight-based doses; 5 days of 1000mg (500mg twice daily) for those weighing <60kg and 5 days of 1500mg (1000mg mane, 500mg nocte) for those weighing ≥60kg
  Arms: Intervention arm

SUMMARY:
This study aims to investigate the effect of metformin as host-directed therapy in obese/overweight patients with dengue

Primary Objective

To evaluate the safety and tolerability of metformin in obese/overweight young adults and children with dengue

Secondary Objectives

* To assess the effect of metformin therapy in obese/overweight patients with dengue on physiological, clinical and virological parameters
* To assess the immunomodulation effects of metformin therapy in obese/overweight patients with dengue
* To assess difference in gene expression between treatment group compared to non-treatment population

DETAILED DESCRIPTION:
This is an open-label safety and tolerability study investigating the effects of five days of metformin treatment. The metformin therapy will be given to eligible participants admitted to the Hospital for Tropical Diseases (HTD) in Ho Chi Minh City, Vietnam. The 60 patients receiving metformin intervention will be compared to 60 age-matched overweight or obese controls, who get the standard supportive treatment only.

The intervention will be conducted in two phases, with a dose escalation. In the initial phase (cohort 1), five young adults (16-30 years) and five children (age 10-16 years) with body mass index (BMI) >25 kg/m2 (BMI-for-age >1 standard deviation - SD) will be provided with a low dose of metformin once daily at 850mg and 500mg respectively. A Data Monitoring Committee (DMC) review will take place after day 5 data is fully available for the first ten patients enrolled in cohort 1. If the five-day safety and clinical data of cohort 1 show no safety concerns, the study will progress to the second phase (cohort 2). This will include 25 adults and 25 children, who will be given a weight-based dose of metformin; 1000mg (500mg twice daily) for participants with weight < 60kg, and 1500mg (1000mg mane, 500mg nocte) for those ≥ 60kg.

Patients that are admitted to the HTD within 72 hours of fever, with clinical suspicion of dengue, will be invited to participate in the trial. After giving consent, patients will be screened for their eligibility to commence treatment with the trial drug. Blood samples will be collected to test for NS1, pregnancy (in all female patients), and AST, ALT and creatinine levels. Glucose and lactate levels will be measured using point-of-care (POC) tests.

All patients will be asked to come back for a final FU visit at around 21-28 days after the onset of fever.

Details of all AEs and SAEs will be recorded on specific forms, together with an assessment as to whether the events are likely to have been related to any treatment received. All SAEs will be reported promptly to the DMC and ECs according to policy. In cases of discontinuation due to AEs, participants will be followed up until the events have resolved or stabilized.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 10 years to ≤ 30 years of age,
* Clinical diagnosis of dengue (based on WHO 2009 Dengue: Guidelines for Diagnosis, Treatment, Prevention and Control/Vietnam Ministry of Health 2019: Guidelines for Dengue Diagnosis, treatment and prevention)
* Positive NS1 rapid test
* ≤ 3 days (≤ 72 hours) of fever
* BMI > 25 Kg/m2 (or BMI-for-age > 1 SD);
* Written informed consent or assent to participate in the study
* Agree to come back for follow up visit around day 21-28 of illness (maximum 1 month)

Exclusion Criteria:

* In all female patients: Pregnancy Localizing features suggesting an alternative diagnosis, e.g. pneumonia, otitis etc.
* History of hypersensitivity to metformin
* Severe infection, including: (1) severe dengue (dengue shock syndrome, severe haemorrhage, severe organ impairment) (2) central nervous system infection, or (3) septicaemia etc…
* Baseline lactate level > 2.0 mmol/L
* Baseline glucose level < 3.9 mmol/L OR < 70 mg/dL
* Already taking metformin or any other regular hypoglycaemic agents, eg. insulin
* Significant diarrhoea and/or vomiting (> 3 episodes in 24 hours)
* Have acute or chronic renal impairment (baseline GFR < 30ml/min)
* Liver impairment (baseline AST and ALT > 250 U/L)
* Being treated for heart failure or have had a recent heart attack (in the last year)
* Taking any drug with significant interaction with metformin
* The study physician judges that the patient is unlikely to attend follow up visit at around 3-4 weeks after fever onset - e.g. due to long travelling distance from the clinic

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to 30 days after enrollment
  Number of severe clinical symptoms and signs, including severe diarrhoea (defined as >5 episodes watery stool/day), severe vomiting (>=3 episodes separated by 15 minutes/24 hours), severe abdominal pain and laboratory markers of severity including -Hypoglycaemia defined as glucose <3.9 mmol/l, Hyperlactatemia (lactate >3 mmol/l), ALT/AST >400 U/l

SECONDARY OUTCOMES:
Fever clearance time | Up to 7 days after enrollment
  Time to temperature <37.5 for 2 consecutive days
Platelet nadir | Up to 7 days after enrollment
  Lowest platelet count recorded during admission
Percentage increase in hematocrit from baseline | Up to 30 days after enrollment
  Percentage increase will be calculated from peak result to baseline (baseline is follow-up time-point)
Percentage change in endothelial and lipid-inflammatory parameters | Up to 30 days after enrollment
  Percentage change in parameters such as: VCAM1, ICAM1, leptin, adiponectin, LDL, AMPK levels will be calculated from peak result to baseline (follow-up time-point)
Changes in virological parameters | Up to 7 days after enrollment
  Area under the curve (AUC) of the serial measurements during days 3 - 6 (log10-transformed), time from enrollment to the first undetectable viraemia, or the first negative NS1 measurement will be compared
Changes in number of immune cells | Up to 30 days after enrollment
  Phenotyping CD8/4+T cell and NK cell and T cell exhaustion markers will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Yacoub, PhD. MD, Principal Investigator — University of Oxford, UK
Locations (1):
- Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data of this study may be requested for publication by journals. Sharing anonymised data with future similar/suitable studies will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be shared with any other person/organisation.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Do LM, Tran TK, Eriksson B, Petzold M, Nguyen CT, Ascher H. Preschool overweight and obesity in urban and rural Vietnam: differences in prevalence and associated factors. Glob Health Action. 2015 Oct 8;8:28615. doi: 10.3402/gha.v8.28615. eCollection 2015. PMID 26452338
- [Background] Dieu HT, Dibley MJ, Sibbritt DW, Hanh TT. Trends in overweight and obesity in pre-school children in urban areas of Ho Chi Minh City, Vietnam, from 2002 to 2005. Public Health Nutr. 2009 May;12(5):702-9. doi: 10.1017/S1368980008003017. Epub 2008 Jul 29. PMID 18664311
- [Background] Nguyen PV, Hong TK, Hoang T, Nguyen DT, Robert AR. High prevalence of overweight among adolescents in Ho Chi Minh City, Vietnam. BMC Public Health. 2013 Feb 15;13:141. doi: 10.1186/1471-2458-13-141. PMID 23414441
- [Background] Zulkipli MS, Dahlui M, Jamil N, Peramalah D, Wai HVC, Bulgiba A, Rampal S. The association between obesity and dengue severity among pediatric patients: A systematic review and meta-analysis. PLoS Negl Trop Dis. 2018 Feb 7;12(2):e0006263. doi: 10.1371/journal.pntd.0006263. eCollection 2018 Feb. PMID 29415036
- [Background] Harris K, Smith L. Safety and efficacy of metformin in patients with type 2 diabetes mellitus and chronic hepatitis C. Ann Pharmacother. 2013 Oct;47(10):1348-52. doi: 10.1177/1060028013503108. PMID 24259699
- [Background] Doyle MA, Singer J, Lee T, Muir M, Cooper C. Improving treatment and liver fibrosis outcomes with metformin in HCV-HIV co-infected and HCV mono-infected patients with insulin resistance: study protocol for a randomized controlled trial. Trials. 2016 Jul 20;17(1):331. doi: 10.1186/s13063-016-1454-6. PMID 27439433
- [Background] Htun HL, Yeo TW, Tam CC, Pang J, Leo YS, Lye DC. Metformin Use and Severe Dengue in Diabetic Adults. Sci Rep. 2018 Feb 20;8(1):3344. doi: 10.1038/s41598-018-21612-6. PMID 29463812
- [Background] Khan IM, Malik BR, Randhawa FA, Butt NF, Malik U, Hamid S. Comparison of metformin and pioglitazone in achieving sustained virological response in chronic hepatitis C patients with insulin resistance: A quasi-experimental study. J Pak Med Assoc. 2017 Dec;67(12):1848-1852. PMID 29256528
- [Background] Padmapriyadarsini C, Bhavani PK, Natrajan M, Ponnuraja C, Kumar H, Gomathy SN, Guleria R, Jawahar SM, Singh M, Balganesh T, Swaminathan S. Evaluation of metformin in combination with rifampicin containing antituberculosis therapy in patients with new, smear-positive pulmonary tuberculosis (METRIF): study protocol for a randomised clinical trial. BMJ Open. 2019 Mar 1;9(3):e024363. doi: 10.1136/bmjopen-2018-024363. PMID 30826761
- [Background] Kay JP, Alemzadeh R, Langley G, D'Angelo L, Smith P, Holshouser S. Beneficial effects of metformin in normoglycemic morbidly obese adolescents. Metabolism. 2001 Dec;50(12):1457-61. doi: 10.1053/meta.2001.28078. PMID 11735093
- [Background] Pastor-Villaescusa B, Canete MD, Villarraso-Caballero J, et al. Metformin for Obesity in Prepubertal and Pubertal Children: A Randomized Controlled Trial. Pediatrics. 2017;140 (1):e20164285. Pediatrics. 2017 Nov;140(5):e20172555. doi: 10.1542/peds.2017-2555. No abstract available. PMID 29089408
- [Background] Soto-Acosta R, Bautista-Carbajal P, Cervantes-Salazar M, Angel-Ambrocio AH, Del Angel RM. DENV up-regulates the HMG-CoA reductase activity through the impairment of AMPK phosphorylation: A potential antiviral target. PLoS Pathog. 2017 Apr 6;13(4):e1006257. doi: 10.1371/journal.ppat.1006257. eCollection 2017 Apr. PMID 28384260
- [Derived] Minh Nguyen N, Thi Hoai Tam D, Quang Chanh H, Trung Trieu H, Thi Xuan Chau N, Thanh Van N, Thanh Phong N, Thi Tam C, Thi Hong Lan N, Thi Hue Tai L, Thi Cam Huong N, Thi Ngoc Thuan L, Van Hao N, Tu Qui P, Thi Dong Vien T, Thi Hai Men P, Thi Thuy Hoa H, Vinh Tho P, Thi Le Duyen H, Tran Thuy V, Dang Trong T, Tan Thanh Kieu N, McBride A, Kestelyn E, Geskus RB, Lam Vuong N, Yacoub S. Safety and tolerability of metformin in overweight and obese patients with dengue: An open-label clinical trial (MeDO). PLoS Negl Trop Dis. 2025 Jul 1;19(7):e0013281. doi: 10.1371/journal.pntd.0013281. eCollection 2025 Jul. PMID 40591696
- [Derived] Nguyen NM, Chanh HQ, Tam DTH, Vuong NL, Chau NTX, Chau NVV, Phong NT, Trieu HT, Luong Thi Hue T, Cao Thi T, Dinh The T, Duyen HTL, Van NTT, Nguyen Than Ha Q, Rivino L, Gallagher P, Jones NK, Geskus RB, Kestelyn E, Yacoub S. Metformin as adjunctive therapy for dengue in overweight and obese patients: a protocol for an open-label clinical trial (MeDO). Wellcome Open Res. 2021 Feb 8;5:160. doi: 10.12688/wellcomeopenres.16053.2. eCollection 2020. PMID 33083561